CLINICAL TRIAL: NCT04859478
Title: Venous Phade Dual Energy Computed Tomography in Patients Suspected for Pulmonary Embolism: Diagnostic Accuracy and Evaluation of Incidental Findings.
Brief Title: Venous Phase Dual Energy CT in Patients Suspected for Pulmonary Embolism.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Yecatarina Zincuk Rohde, MD, MD, Copenhagen University Hospital at Herlev
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-20035522
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Embolus/Emboli; Thromboembolism, Pulmonary
Keywords: CT; CTPA; Computed tomography; Computed tomography pulmonary angiography; Dual energy; Spectral; Sensitivity; Incidental findings; Iodine mapping; Radiology; Imaging; Diagnostic accuracy
MeSH Terms: conditions — Pulmonary Embolism; Embolism; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All eligible patients (Other): All patients undergo the same CT protocol in addition to standard care.
  Interventions: Diagnostic Test: Dual energy / spectral portal venous chest computed tomography

INTERVENTIONS:
Diagnostic Test: Dual energy / spectral portal venous chest computed tomography — Each patient undergoes an additional dual energy / spectral chest CT in addition to standard care CTPA. The intervention is performed immediately after standard care CTPA.

SUMMARY:
Venous phase spectral or dual energy (DE) chest computed tomography (CT) in patients with suspected pulmonary embolism (PE) compared to standard computed tomography pulmonary angiography (CTPA): sensitivity, evaluation of iodine mapping and incidental findings.

DETAILED DESCRIPTION:
Background/rationale: DE CTPA provides additional anatomical and functional information in the investigation of PE, especially in regards of iodine uptake in pulmonary vasculature and lung parenchyma. Postprocessing techniques improve visualisation of low concentrations of iodine contrast media.This has shown potential in reducing the amount of contrast media, salvaging scans with suboptimal contrast enhancement and for improving visualisation of incidental pulmonary embolisms in portal venous chest CT scans. Other significant DE postprocessing techniques include the substraction of iodine, creating virtual non-contrast images in addition to the dual energy. This technique has proven useful in evaluation of different thoracic and abdominal parenchymal lesions.

Objective: To evaluate sensitivity of chest DECT in portal venous phase in the diagnosis of PE compared to standard care DE CTPA. Furthermore, the prevalence and management of incidental findings will be evaluated.

Design: Patients enrolled in this study will undergo a venous phase chest DE CT in addition to standard care DE CTPA. The two scans will be performed consecutively using the same contrast media bolus. Standard DE reconstructions of all scans will be obtained for radiological evaluation and reporting in regards of suspected PE.

Both scans with standard DE reconstructions will be available for clinical evaluation and patient care in the standard care AGFA PACS system. Radiological reading and reporting will be performed as usual in the clinical setting.

For research purposes, additional post-processing procedures may be performed by the readers in Philips IntelliSpace Portal or Siemens Syngo.via depending on the scanner applied. The standard CTPA will be interpreted by a thoracic radiologist and used as reference. The corresponding portal venous chest CT will be interpreted individually by two other certified radiologists in order to avoid recall bias. In case of disagreement in the venous chest CT, an independent radiologist not elsewhere involved will be consulted. If a PE detected on the portal venous scan is not detected on the reference CTPA, the reference reader will re-evaluate the CTPA.

Patient characteristics, clinical information, radiation dose, contrast media, clinical diagnosis, incidental findings and recommendations of further clinical management according to clinical guidelines will be recorded in a secure web-based database.

Study population: Patients aged ≥50 with suspected pulmonary embolism who are having performed a standard care CTPA.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected for pulmonary embolism undergoing a computed tomography pulmonary angiography
* Minimum age 50 years

Exclusion Criteria:

* Temporarily or permanently incompetent patient not able to give informed consent
* No informed consent obtained for other reasons
* Allergic to iodine based contrast media
* Impaired renal function
* Patients with thyreotoxicosis
* Non-diagnostic quality of computed tomography images

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | through study completion, approx. of 1 year
  Per patient sensitivity of portal venous phase chest DECT in diagnosing PE compared to the corresponding reference CTPA
Specificity | through study completion, approx. 1 year
  Per patient specificity of portal venous phase chest DECT in diagnosing PE compared to the corresponding reference CTPA

SECONDARY OUTCOMES:
Sensitivity | through study completion, approx. of 1 year
  Lobe and segment based sensitivity of portal venous phase chest DECT in diagnosing PE compared to the corresponding reference CTPA
Specificity | through study completion, approx. of 1 year
  Lobe and segment based specificicty of portal venous phase chest DECT in diagnosing PE compared to the corresponding reference CTPA
Incidental findings | through study completion, approx. of 1 year
  Evaluation and management of incidental findings in portal venous phase chest CT compared to standard care CTPA.
Iodine mapping | through study completion, approx. of 1 year
  Comparison of perfusion defects on iodine mapping between portal venous chest CT and CTPA. Descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Yecatarina Z Rohde, MD, Principal Investigator — Copenhagen University Herlev Hospital
Locations (2):
- Denmark (2):
  - Copenhagen University Gentofte Hospital, Copenhagen, Hellerup
  - Copenhagen University Hospital, Herlev Hospital, Copenhagen, Herlev

IPD SHARING:
Plan to Share IPD: No